CLINICAL TRIAL: NCT00360516
Title: Paleolithic Diets, Exercise Physiology and Metabolism
Brief Title: Paleolithic Diet and Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: GCRC, UCSF
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H8748-27380-02
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Diet
Keywords: healthy volunteers
MeSH Terms: interventions — Metabolic Networks and Pathways; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: metabolic (nutrient controlled) diet — metabolic (nutrient controlled) diet

SUMMARY:
If eating a "Paleolithic" diet helps improve these diseases, this would be the first step in both improving people's health as they get older as well as contributing to future national dietary guidelines for Americans.

DETAILED DESCRIPTION:
Because genetic evolutionary changes occur slowly in Homo sapiens, and because the traditional diet of Homo sapiens underwent dramatic changes within recent times, modern humans are better physiologically adapted to a diet similar to the one their hominid ancestors evolved on than to the diet typical of modern industrialized societies. The investigators developed a computational model to estimate the net acid load of diets from the nutrient composition of the diet's component ingredients, and suggest that the majority of these hominid diets yield a negative net acid load (that is, yield a net base load), in addition to being low in sodium chloride, high in potassium-containing fruits and vegetables, and low in saturated fats, with the majority of the non-animal-source calories coming from fruits and vegetables, not from acid-producing grains, separated fats and oils, starches and refined sugars. According to paleonutritionists, Homo sapiens' recent switch from their ancestral Paleolithic-type diet to the modern Western diet has contributed in a major way to so-called age-related diseases of civilization. The investigators hypothesize and will test whether:

1. consuming a high-potassium, low-sodium, net base-producing "Paleolithic-type" diet, even in the short term, has detectable beneficial effects on cardiovascular physiology, serum lipid profiles, insulin sensitivity, and exercise performance; and
2. their computational model predicts the measured negative net acid loads of a net base-producing "Paleolithic-type" diet, using steady-state values of renal net acid excretion as the measure of the diet net acid load (a.k.a., net endogenous acid production), which will be of value in constructing net-base producing diets for modern consumption.

The long term complications of the combination of high blood pressure, high blood sugar and high fat and cholesterol levels, sometimes called the "metabolic syndrome", has been termed the number one medical problem in modern society today. If eating a "Paleolithic" diet helps improve these diseases, this would be the first step in both improving people's health as they get older as well as contributing to future national dietary guidelines for Americans.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and <= 55 years
* On no medications
* Body mass index (BMI) between 18 and 29.9 kg/m2
* Normal renal and hepatic function
* Subjects who report moderate intensity exercising <= three times a week for 30 minutes or less, who then qualify by exercise testing with a VO2max at or below age- and gender-matched controls

Exclusion Criteria:

* Subjects who must follow a specific diet
* Subjects on any daily medications
* Subjects unwilling to follow the diet specified
* Subjects unable to do the exercise testing
* Pregnant women
* Subjects who are unable to understand the consent form.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
validation of algorithm to predict diet net acid load | 1year
  measuring 24-hour net acid and comparing this to the estimated diet acid load using one of several algorithms

SECONDARY OUTCOMES:
effects of a "Paleolithic" diet on exercise capacity, vascular reactivity, lactate production during exercise, glucose and lipid profiles and | 1 year
  measuring VO2max, CO, BAR,

CONTACTS AND LOCATIONS:
Overall Officials: Lynda A Frassetto, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF 505 Parnassus Ave, San Francisco, California, United States

REFERENCES:
- [Background] Sebastian A, Frassetto LA, Sellmeyer DE, Merriam RL, Morris RC Jr. Estimation of the net acid load of the diet of ancestral preagricultural Homo sapiens and their hominid ancestors. Am J Clin Nutr. 2002 Dec;76(6):1308-16. doi: 10.1093/ajcn/76.6.1308. PMID 12450898
- [Background] Frassetto L, Morris RC Jr, Sellmeyer DE, Todd K, Sebastian A. Diet, evolution and aging--the pathophysiologic effects of the post-agricultural inversion of the potassium-to-sodium and base-to-chloride ratios in the human diet. Eur J Nutr. 2001 Oct;40(5):200-13. doi: 10.1007/s394-001-8347-4. PMID 11842945